CLINICAL TRIAL: NCT06637280
Title: HFNC Versus Conventional Nasal Cannula During EBUS Procedure: a Randomised Controlled Trial
Brief Title: High - Flow Nasal Cannula Versus Conventional Nasal Cannula During Endobronchial Ultrasound Procedure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Collaborators: National and Kapodistrian University of Athens (Other); Clinical Hospital Centre Zagreb (Other); Universidade Nova de Lisboa (Other)
Responsible Party: Principal Investigator, Aleš Rozman, MD, PhD, specialist for chest diseases, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0120-294/2023/3
Record Dates: First submitted 2024-09-29; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Hypoxemia During EBUS Bronchoscopy
Keywords: EBUS bronchoscopy; high - flow nasal cannula; oxygenation; desaturation; oxygen supplementation

STUDY DESIGN:
Intervention Model Description: randomised, prospective
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard nasal cannula 6l/min, 100% O2 (Active Comparator): Standard procedure during EBUS bronchoscopy
  Interventions: Device: Standard nasal cannula
- High - flow nasal cannula 60l/min, 45% O2 (Experimental): The new method
  Interventions: Device: High - flow nasal cannula

INTERVENTIONS:
Device: High - flow nasal cannula — High flow nasal cannula (HFNC), a device first introduced in neonates and pediatric care, is currently used in a wide range of indications in adult respiratory and critical care medicine (5-7). It is a relatively new method in bronchoscopy with several notable theoretical advantages over low flow oxygen via conventional nasal cannula (CNC):
  * High flow up to 60 liters per minute ensures a more stable FiO2 and better matches the increased patient's inspiratory flow
  * High flow generates a small positive expiratory airway pressure (up to 5 cm H2O) which could stabilize the upper airways during sedation and have a beneficial effect in the lower airways
  * High flow reduces dead space in the upper airways and increases alveolar ventilation.
  Arms: High - flow nasal cannula 60l/min, 45% O2
Device: Standard nasal cannula — Standard method for supplementing oxygen during EBUS bronchoscopy
  Arms: Standard nasal cannula 6l/min, 100% O2

SUMMARY:
EBUS bronchoscopy is performed in most centers under local anesthesia and moderate sedation. Both the bronchoscopy itself and the sedation can lead to decreased ventilation and a drop in oxygen saturation in the body. Typically, oxygen is administered during the procedure via a nasal cannula at a flow rate of 6l/min. The aim of the study is to compare a new method - a nasal cannula with high flow - to the standard cannula. The primary objective is to demonstrate that the new method is more effective at preventing desaturation during the procedure. Patients will be randomized into two groups before bronchoscopy and monitored. The bronchoscopy will be performed in the same way for both groups. The only difference between the groups will be in the method of oxygen administration during EBUS bronchoscopy.

DETAILED DESCRIPTION:
Introduction

1. EBUS - bronchoscopy From a physiological point of view bronchoscopy is an introduction of a foreign body into the airway. Response mechanisms include laryngospasm, bronchospasm, cough, increased secretion of bronchial mucus and reduced depth of breathing. Sympathetic response with increased heart rate and blood pressure is common even before the procedure, while the patient is being prepared on the examination table. The bronchoscope occupies 10 to 15% of the cross-sectional area in the major airways and increases air flow resistance. Suction applied during the procedure causes air stealing through the working channel of the bronchoscope which reduces end inspiratory and expiratory volumes leading to alveolar de-recruitment with increased intrapulmonary shunting consequently.

   EBUS bronchoscopy is associated with prolonged procedure time, increased airway contact, a thicker instrument, and multiple needle punctures through the tracheal and/or bronchial wall. All these factors cause additional stress to the patient and require additional local anesthesia and deeper level of sedation.
2. Sedation Although topical anesthesia of the upper airways, vocal cords, trachea, and bronchi enables a tolerable bronchoscopic procedure, a moderate level of sedation during bronchoscopy is currently the golden standard. Use of sedation facilitates the passage through the vocal cords, inhibits airway protective reflexes and increases patient safety (2,3). In combination with physiological responses to bronchoscopy which increase oxygen demand, sedatives used during bronchoscopy reduce respiratory drive and further compromise patients, especially those with chronic diseases. When it occurs, hypoxemia can induce periprocedural arrythmias and ischemia therefore should be generally avoided and, if encountered, must be reverted quickly (4). An oxygenation strategy with appropriate oxygen supplementation is therefore required during most bronchoscopic procedures.
3. Oxygen supplementation Low flow oxygen up to 6 liters per minute applied through a nasal catheter is the most often used method for oxygen supplementation during flexible bronchoscopy. Inspired oxygen fraction (FiO2) can reach up to 45% but cannot be reliably predicted and may not be enough in all cases.

   High flow nasal cannula (HFNC), a device first introduced in neonates and pediatric care, is currently used in a wide range of indications in adult respiratory and critical care medicine (5-7). It is a relatively new method in bronchoscopy with several notable theoretical advantages over low flow oxygen via conventional nasal cannula (CNC):
   * High flow up to 60 liters per minute ensures a more stable FiO2 and better matches the increased patient's inspiratory flow
   * High flow generates a small positive expiratory airway pressure (up to 5 cm H2O) which could stabilize the upper airways during sedation and have a beneficial effect in the lower airways
   * High flow reduces dead space in the upper airways and increases alveolar ventilation.

   CPAP and NIV can provide similar beneficial effects, but their use is challenging because they require a close-fitting facial mask which limits the use of a bronchoscope, aspiration of secretions from the upper airways, pharynx, or oral cavity and expectoration of sputum.
4. Previous studies on HFNC

   A recent meta-analysis which included six randomized controlled trials found that patients who underwent bronchoscopy with the use of HFNC experienced less hypoxemic events and desaturations, had fewer procedural interruptions and pneumothorax compared to patients supplemented with CNC (10). The three studies which evaluated HFNC during EBUS all showed that HFNC is more effective than CNC during the procedure and that HFNC can be considered an alternative to CNC. However, the studies had several important limitations such as a low number of patients included with a historical control (Takakuwa O et al), a large difference in FiO2 between trial groups (2L/min in the CNC vs. 100% FiO2 and 70L/min flow rate in the HFNC group) (Irfan et al) and lack of assessment of CO2 levels during the procedure (Ulcar et al). Nevertheless, conclusions suggested that HFNC is sufficiently safe and provides adequate oxygenation for most of bronchoscopy examinations including EBUS (8,9).
5. Study questions

Our hypothesis is that HFNC provides better control over hypoxemia during EBUS-TBNA procedure than CNC. The primary outcome of the study is therefore proportion of patients with successfully controlled hypoxemia during EBUS TBNA in each arm. Secondary outcomes are incidence of complications in each arm (number of hypoxemic events, mean lowest oxygen saturation during procedure, average saturation, drop in saturation, pulse rate, blood pressure, incidence of arrhythmia), number of patients who experienced mild, moderate, or severe hypoxemia, number of patients who required escalation of the support and which support is effective, what are risk factors for desaturation.

Methods

1. Study design and study population

   The study is designed as multicenter randomized controlled prospective trial. Study will enroll patients who need EBUS -TBNA procedure with sampling of mediastinal lymph nodes for diagnosis and/or staging.

   Patients will be recruited from four university hospitals in Slovenia, Croatia, Portugal and Greece.

   Study was approved by The National Medical Ethics Committee of the Republic of Slovenia and registered as 0120-294/2023/3.
2. Recruitment, consensus, and randomization

   Bronchoscopy coordinator will screen the scheduled patients and notify study investigator about eligible patients. Study investigator will explain the study to eligible patients and obtain informed consents. Inclusion and exclusion criteria will be checked on the day of examination from the data routinely obtained before procedure, including laboratory data.

   Patients will be randomized in bronchoscopy suite according to allocation group written in sequentially numbered, sealed and opaque envelopes. Envelopes will be prepared by independent statistician on the basis of block randomization with the block size of 4.
3. Bronchoscopy and sedation

   Topical anesthesia with lidocaine will be provided routinely before insertion of the bronchoscope. Patients will be sedated by bedside anesthesiologist by combination of midazolam, fentanyl and propofol. The depth of sedation will be assessed using Modified Observer's Assessment of Alertness / Sedation scale (MOAA/S). The level of sedation will be maintained between 1 and 2 throughout the procedure. Patients will be monitored by BIS monitor for further analysis and comparison.

   The standard group of patients will receive oxygen through double-prong nasal cannula with the oxygen flow set to 6 liters per minute, which corresponds to FiO2 45%. The HFNC group will receive mixture of oxygen and air at FiO2 45% with initial flow of 60 liters per minute pre-warmed to 37 degrees of Celsius. Nasal cannula will be chosen according to the patient's face size. Before procedure, patients from both groups will be tested with HFNC with the flow of 60 l/min if they are able tolerate it.

   EBUS bronchoscope will be inserted through the oral bite block by experienced bronchoscopist and the whole procedure will be conducted according to ERS recommendations. After systematical evaluation of mediastinal and hilar lymph nodes, EBUS TBNA's will be performed according to the individual procedure plan.

   Patients will be monitored by continuous pulse oximetry, periodical blood pressure measurements, ECG and BIS.
4. Hypoxemia escalation protocol, complications, and termination criteria

Oxygen will be delivered to the patient according to the allocation group (6l/min O2 CNC or 45% FiO2 60 l/min HFNC). If desaturation occurs, defined as SpO2<90% for more than 10s the patients will be approached according to the escalation protocol (Figure 1):

1. jaw thrust maneuver
2. patients in CNC group will be switched to 45% FiO2 60 l/min HFNC
3. patients with 45% FiO2 60 l/min HFNC will be switched to 100% FiO2
4. patients with HFNC failure will be switched to advanced respiratory support (balloon ventilation, laryngeal mask, intubation, reversal of sedation)

   In the case of moderate hypoxemia there will be temporal suspension of the bronchoscopy but in the case of severe hypoxemia the termination of the procedure will be considered if there is no immediate improvement after escalation of ventilatory support.

   Procedure will be terminated also in the case of other severe adverse events as are hemodynamic instability, myocardial ischemia, or pneumothorax. Resuscitation equipment will be prepared on dedicated medical cart inside the bronchoscopy suite. Any patient with adverse event will be monitored until complete recovery (Alderete score 9 or more).

   Complications, relevant to the decisions and study outcomes are defined as (1):
   * Desaturation <90% for more than 10s
   * Moderate desaturation 75%<= SpO2 <90% less than 60s
   * Severe desaturation <75% or 75%<= SpO2 <90% more than 60s
   * Tachycardia >100 or +25%
   * Bradycardia <50 or -25%
   * Hypertension +25%
   * Hypotension <90mmHg or -25%
5. Data collection

   Demographic data of patients (age, gender, height, weight, BMI, STOP-BANG score, ASA score) and laboratory results (lung function testing) relevant for the study will be collected before the procedure. During and after the procedure, there will be continuous (SpO2, pulse rate, ECG) or periodical (blood pressure) monitoring of vital signs and depth of the sedation (BIS, MOAA/S). The starting point of the procedure T0 is defined as the time immediately prior sedatives are given to the patient. T1 is the time point, where bronchoscope is inserted and Tend is the end of the procedure, when bronchoscope is withdrawn. Venous blood for pCO2 analysis will be drawn at T0 (on the procedure table before sedation) and at Tend (withdrawal of the bronchoscope).

   Timing and duration of desaturation, the lowest SpO2 and all treatment escalations will be recorded as well as other possible complications.
6. Sample size

   The protocol is designed to show a superiority of HFNC over CNC. According to pulled data in recently published meta-analysis we expect a 12% desaturation rate in the HFNC group and a 34% desaturation rate in CNC group. The sample size should be 112 with a confidence level (alpha) of 95%, power (1-beta) of 80%. With expected drop out of 25% the final number of included participants is set to 150. A web-based application was used for sample size calculation (https://clincalc.com/stats/samplesize.aspx).
7. Statistical analysis

   Data will be collected in specially designed case report formulars (CRF) and analyzed by GraphPad Prism 9.5. software (Boston, MA). Categorical variables will be presented as percentages and analyzed by chi-square test. Numerical variables will be presented as mean and standard deviation or median and ranges. Distribution will be tested by the Kolmogorov - Smirnov test and further analysis performed by t-test or Mann Whitney test depending on normality of distribution. Two-sided p-value will be regarded as statistically significant if < 0,05.
8. Patient and public involvement

Patients and public were not involved in the study design.

References:

1. Mason KP, Green SM, Piacevoli Q; International Sedation Task Force. Adverse event reporting tool to standardize the reporting and tracking of adverse events during procedural sedation: a consensus document from the World SIVA International Sedation Task Force. Br J Anaesth. 2012 Jan;108(1):13-20. doi: 10.1093/bja/aer407. PMID: 22157446.
2. Sazak H, Tunç M, Alagöz A, Pehlivanoğ Lu P, Demirci NY, Alıcı İO, et al. Assessment of perianesthesic data in subjects undergoing endobronchial ultrasound-guided transbronchial needle aspiration. Respir Care. 2015;60(4):567-76.
3. Douglas N, Ng I, Nazeem F, Lee K, Mezzavia P, Krieser R, et al. A randomised controlled trial comparing high-flow nasal oxygen with standard management for conscious sedation during bronchoscopy. Anaesthesia. 2018;73(2):169-76.
4. Du Rand IA, Blaikley J, Booton R, Chaudhuri N, Gupta V, Khalid S, et al. British Thoracic Society guideline for diagnostic flexible bronchoscopy in adults: accredited by NICE. Thorax. 2013 Aug;68 Suppl 1:i1-44.
5. Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-Flow Nasal Cannulae in the Management of Apnea of Prematurity: A Comparison With Conventional Nasal Continuous Positive Airway Pressure. Pediatrics [Internet]. 2001 May 1;107(5):1081-3. Available from: https://doi.org/10.1542/peds.107.5.1081
6. Roca O, Riera J, Torres F, Masclans JR. High-Flow Oxygen Therapy in Acute Respiratory Failure. Respir Care [Internet]. 2010 Apr 1;55(4):408 LP - 413. Available from: http://rc.rcjournal.com/content/55/4/408.abstract
7. Nishimura M. High-Flow Nasal Cannula Oxygen Therapy Devices. Respir Care [Internet]. 2019 Jun 1;64(6):735 LP - 742. Available from: http://rc.rcjournal.com/content/64/6/735.abstract
8. Takakuwa O, Oguri T, Asano T, Fukuda S, Kanemitsu Y, Uemura T, et al. Prevention of hypoxemia during endobronchial ultrasound-guided transbronchial needle aspiration: Usefulness of high-flow nasal cannula. Respir Investig. 2018;56(5):418-23.
9. Irfan M, Ahmed M, Breen D. Assessment of High Flow Nasal Cannula Oxygenation in Endobronchial Ultrasound Bronchoscopy: A Randomized Controlled Trial. J Bronchol Interv Pulmonol. 2021;28(2):130-7.
10. Su C-L, Chiang L-L, Tam K-W, Chen T-T, Hu M-C (2021) High-flow nasal cannula for reducing hypoxemic events in patients undergoing bronchoscopy: A systematic review and meta- analysis of randomized trials. PLoS ONE 16(12): e0260716. https://doi.org/10.1371/journal. pone.0260716

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years, ASA I - III, with normal pre-procedural pO2 (> 8.0 kPa) and pCO2 (< 6.7 kPa) levels without oxygen supplementation

Exclusion Criteria:

* - Patient refuses to participate in the study
* Contraindication for topical anesthesia, iv sedation, or bronchoscopy
* Pregnancy
* Contraindication for HFNC including nasopharyngeal obstruction and blockage
* Patient unable to tolerate HFNC 60l/min (tested before the procedure)
* Procedure shorter than 10 min
* Less than 3 EBUS-TBNAs performed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of desaturations during EBUS bronchoscopy | From beginning of EBUS bronchoscopy until the end of the procedure + 10 minutes
  * Desaturation <90% for more than 10 seconds
  * Moderate desaturation 75% <= SpO2 <90% less than 60 seconds
  * Severe desaturation <75% or 75% <= SpO2 <90% more than 60 seconds

CONTACTS AND LOCATIONS:
Locations (4):
- University Hospital Centre Zagreb - Jordanovac, Zagreb, City of Zagreb, Croatia
- National and Kapodistrian University of Athens, Athens, Athens, Greece
- Clinica Universitaria de Pneumologia, Hospital de Santa Maria, Lisbon, Lisbon District, Portugal
- University Clinic Golnik, Golnik, Golnik, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Publication in a peer - reviewed journal
Supporting Information: CSR
Time Frame: In 2025
Access Criteria: open access journal preferably